CLINICAL TRIAL: NCT00806715
Title: Impact of Iron Overload in Pediatric Patients Undergoing Stem Cell Transplantation
Brief Title: Iron Overload in Stem Cell Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Lance Armstrong Foundation (Other)
Responsible Party: Principal Investigator, Deborah Chirnomas, Instructor, Boston Children's Hospital
Other Study IDs: DFCI 07-004
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2011-06

CONDITIONS: Iron Overload
Keywords: hemochromatosis; Iron overload; Stem cell transplant; Pediatrics; Pediatric Stem cell transplant
MeSH Terms: conditions — Iron Overload; Hemochromatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood specimens.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to examine the impact of iron overload in patients undergoing a bone marrow transplant. We believe that the iron status in these patients is associated with complications for transplant survivors. We will examine the iron status in these patients by MRI and by screening for mutations in genes known to cause iron overload. We will also determine the levels of hepcidin (a hormone produced in the liver that appears to regulate iron homeostasis) from blood and urine.

ELIGIBILITY:
1. Undergoing allogeneic HSCT for malignant or non-malignant conditions
2. Age greater than or equal to 5 years
3. Able to undergo MRI without a need for general anesthesia
4. No metal implants
5. Signed informed consent (by parent if patient is less than 18 years old, or by patient, if he or she is greater than 18 years old).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children undergoing allogeneic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Hepatic iron content as measured by R2 MRI. | Pre-HSCT and Day 100

SECONDARY OUTCOMES:
Genetic determinants of iron overload- HFE status. | Pre-HSCT

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States